CLINICAL TRIAL: NCT04174157
Title: A Prospective, Long-Term Registry of Patients With a Diagnosis of Spinal Muscular Atrophy (SMA)
Brief Title: Registry of Patients With a Diagnosis of Spinal Muscular Atrophy (SMA)
Status: Recruiting | Type: Observational
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Other Study IDs: COAV101A12001
Expanded Access: NCT03955679 (Approved for marketing)
Record Dates: First submitted 2019-09-12; First posted 2019-11-22 (Actual); Last update posted 2025-01-31 (Actual); Status verified 2025-01

CONDITIONS: Spinal Muscular Atrophy (SMA)
MeSH Terms: conditions — Muscular Atrophy, Spinal | interventions — Zolgensma

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 15 Years
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Prospective observational registry: This is a prospective, multi center, multinational, non-interventional observational registry.
  Interventions: Other: Prospective observational registry; Drug: Zolgensma

INTERVENTIONS:
Other: Prospective observational registry — This prospective observational registry will assess long-term outcomes of patients with a diagnosis of SMA.
Drug: Zolgensma — Zolgensma will be given to patients as per normal clinical practice and clinical care will not be mandated by the protocol. As such, the decision to prescribe Zolgensma is separate from the decision to include the patient in this study

SUMMARY:
Spinal muscular atrophy (SMA) is a neurogenetic disorder caused by a loss or mutation in the survival motor neuron 1 gene (SMN1) on chromosome 5q13, which leads to reduced SMN protein levels and a selective dysfunction of motor neurons. SMA is an autosomal recessive, early childhood disease with an incidence of 1:10,000 live births. SMA is the leading cause of infant mortality due to genetic diseases.

The purpose of this registry is to assess the long term outcomes of patients with SMA in the context of advances in treatment options and also to characterize and assess long-term safety and effectiveness of OAV-101.

DETAILED DESCRIPTION:
This is a prospective, multi center, multinational, non-interventional observational study. All patients will be managed according to the clinical site's normal clinical practice, i.e., the diagnostic and clinical treatment/practice process that a clinician chooses according to their clinical judgement for an SMA patient. Clinical care will not be driven by the protocol. No additional visits or investigations will be performed beyond normal clinical practice. Patients will be followed for 15 years from enrolment or until death, whichever is sooner.

ELIGIBILITY:
Inclusion Criteria:

* Patients treated with OAV-101 with a genetically confirmed diagnosis of SMA regardless of the date of diagnosis.
* Appropriate consent/assent has been obtained for participation in the registry

Exclusion Criteria:

- Currently enrolled in an interventional clinical trial involving an investigational medicinal product to treat SMA.

Note: Patients who are participating in a Compassionate Use Program (CUP) for OAV-101 (Zolgensma) such as a Managed Access Program (MAP), an Expanded Access Program (EAP), Single Patient Investigational New Drug (IND) (SPI) or Named Patient Program (NPP) are eligible to enroll in the registry regardless of the date of a genetic or clinical diagnosis of SMA.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study will enroll at least 500 patients with a genetically confirmed diagnosis of SMA. The registry will attempt to enroll all patients treated with OAV-101 in the registry until the end of 2026.
Sampling Method: Non-Probability Sample
Enrollment: 700 (Estimated)
Dates: Start 2018-09-25 (Actual); Primary Completion 2038-06-30 (Estimated); Study Completion 2038-06-30 (Estimated)

PRIMARY OUTCOMES:
Change in probability of survival of all patients with SMA using Kaplan Meier method to estimate | Based on information collected at Baseline and every 6 months through 2 years of follow-up, then annually through 15 years of follow up.
Change from baseline Children's Hospital of Philadelphia Infant Test of Neuromuscular Disorders (CHOP-INTEND) in infants with pre-symptomatic or type I SMA | Baseline and every 6 months through 2 years of follow up, then annually through 15 years of follow up
  CHOP INTEND score ranges from 0 to 64 with higher scores indicating higher motor function
Change from baseline Hammersmith Infant Neurological Examination (HINE) in infants with pre-symptomatic, type I or type II SMA | Baseline and every 6 months through 2 years of follow up, then annually through 15 years of follow up
  HINE score range from 0 to 26 with higher scores indicating more development.
Change from baseline in Hammersmith Functional Motor Scale Expanded (HFMSE) for patients with type II and III SMA | Baseline and every 6months through 2 years of follow up, then annually through 15 years of follow up
  HFMSE score range from 0 to 66 with the higher scores indicating more development.
Incidence of treatment emergent adverse events | Through 15 years of follow up
Incidence of treatment emergent serious adverse events | Through 15 years of follow up
Incidence of treatment emergent adverse events related to therapy | Through 15 years of follow up
Incidence of treatment emergent thrombocytopenia, hepatotoxicity and cardiac adverse events | Through 15 years of follow up

SECONDARY OUTCOMES:
Change from baseline in rates of hospitalization | Baseline and every 6 months through 2 years of follow up, then annually through 15 years of follow up
Change from baseline in Zarit Burden Interview | Baseline and every 6 months through 2 years of follow up, then annually through 15 years of follow up
  Zarit Burden Total Score ranges from 0 to 88. A higher score correlates with higher level of burden.
Change from baseline in PedsQL Patient interview | Baseline and every 6 months through 2 years of follow up, then annually through 15 years of follow up
  PedsQL Total Scale Score is average of all items and ranges from 0 to 100. A higher score correlates with better Health-Related Quality of Life
Change from baseline in PedsQL Parent interview | Baseline and every 6 months through 2 years of follow up, then annually through 15 years of follow up
  PedsQL Total Scale Score is average of all items and ranges from 0 to 100. A higher score correlates with better Health-Related Quality of Life
Change from baseline in percent of patients requiring ventilator support (BiPAP, Endotracheal tube) | : Baseline and every 6 months through 2 years of follow up, then annually through 15 years of follow up
Change from baseline in in percent of patients requiring nutritional support (Gastrostomy Tube, Gastrojejunal tube (GT) with Nissen fundoplication, GT without Nissen fundoplication, Nasogastrictube, Nasojejunaltube or Percutaneous endoscopic gastrostomy) | Baseline and every 6 months through 2 years of follow up, then annually through 15 years of follow up
Change from baseline in in percent of patients requiring mobility device support (Ankle-Foot Orthoses, Supramalleolar Orthosis, Orthotic/shoe inserts, Knee immobilizers, Knee-Ankle-Foot Orthoses , Hand splints, Spinal bracing) | : Baseline and every 6 months through 2 years of follow up, then annually through 15 years of follow up

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (99):
- United States (50):
  - Phoenix Children's Hospital, Phoenix, Arizona
  - Arkansas Children's Hospital, Little Rock, Arkansas
  - Loma Linda University Health, Loma Linda, California
  - Children's Hospital of Los Angeles, Los Angeles, California
  - University of California Los Angeles Health, Los Angeles, California
  - Valley Children's Healthcare, Madera, California
  - Children's Hospital of Orange County, Madera, California
  - University of California Davis Health System, Sacramento, California
  - Rady Children's Hospital San Diego, San Diego, California
  - Children's Hospital Colorado, Aurora, Colorado
  - Connecticut Children's Medical Center, Farmington, Connecticut
  - Yale-New Haven Health System, New Haven, Connecticut
  - Golisano Children's Hospital of Southwest Florida, Fort Myers, Florida
  - Nicklaus Children's Hospital, Miami, Florida
  - Adventist Health System - Florida, Orlando, Florida
  - Jackson South Medical Center, Palmetto Bay, Florida
  - Indiana University Health University Hospital (IUHUH), Indianapolis, Indiana
  - University of Iowa, Iowa City, Iowa
  - University of Kansas Medical Center, Kansas City, Kansas
  - University of Louisville, Louisville, Kentucky
  - University of Minnesota, Minneapolis, Minnesota
  - University of Missouri Health System, Columbia, Missouri
  - Washington University School of Medicine in St. Louis, St Louis, Missouri
  - Atlantic Health System, Morristown, New Jersey
  - University of Rochester Medical Center, Rochester, New York
  - The State University of New York, Stony Brook, New York
  - Duke Health, Durham, North Carolina
  - Akron Children's Hospital, Akron, Ohio
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - University Hospitals, Cleveland, Ohio
  - Nationwide Children's Hospital, Columbus, Ohio
  - Oklahoma University Medical Center, Oklahoma City, Oklahoma
  - Oregon Health and Science University, Portland, Oregon
  - Penn State Hershey, Hershey, Pennsylvania
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Prisma Health, Greenville, South Carolina
  - Methodist Le Bonheur Healthcare, Memphis, Tennessee
  - Child Neurology Consultants of Austin, Austin, Texas
  - Children's Health, Dallas, Texas
  - Cook Children's, Fort Worth, Texas
  - Texas Children's Hospital, Houston, Texas
  - CHRISTUS Health, San Antonio, Texas
  - University of Utah, Salt Lake City, Utah
  - University of Virginia Health System, Charlottesville, Virginia
  - Children's Hospital of The King's Daughters, Norfolk, Virginia
  - Virginia Commonwealth University Health System, Richmond, Virginia
  - Seattle Children's, Seattle, Washington
  - MultiCare Health System, Tacoma, Washington
  - University of Wisconsin, Madison, Wisconsin
  - Children's Hospital of Wisconsin, Milwaukee, Wisconsin
- Greece (4):
  - University General Hospital Attikon, Chaïdári, Athens
  - Penteli Children's Hospital, Pentéli, Attikis
  - St. Sophia Children's Hospital, Thessaloniki
  - General Hospital of Thessaloniki Ippokrateio, Thessaloniki
- Children's University Hospital-UCD School of Medicine Scoil an Leighis, Dublin, Ireland
- Israel (4):
  - Soroka Medical Centre, Beersheba
  - Wolfson Medical Center, Holon
  - Tel-Aviv Sourasky Medical Center, Holon
  - Schneider- Children's Medical Center, Petah Tikva
- Japan (19):
  - Aichi Medical University Hospital, Nagakute-shi, Aichi-ken
  - Fujita Health University Hospital, Toyoake-shi, Aichi-ken
  - Chiba children's Hospital, Chiba, Chiba
  - Kurume University Hospital, Kurume-shi, Fukuoka
  - Gifu Prefectural General Medical Center, Gifu, Gifu
  - Sapporo Medical University Hospital, Sapporo, Hokkaido
  - Kagawa University Hospital, Kita-gun, Kagawa-ken
  - Kanagawa Children's Medical Center, Yokohama, Kanagawa
  - Kumamoto University Hospital, Kumamoto, Kumamoto
  - Miyagi Children's Hospital, Sendai, Miyagi
  - Obihiro Kosei Hospital, Hokkaido, Obihiro-shi
  - Shiga Medical Center for Children, Moriyama-shi, Shiga
  - Hamamatsu University School of Medicine, University Hospital, Hamamatsu, Shizuoka
  - Jichi Medical University Hospital, Shimotsuke-shi, Tochigi
  - Tokyo Medical University Hospital, Shinjuku-ku, Tokyo
  - Center Hospital of the National Center for Global Health and Medicine, Shinjuku-ku, Tokyo
  - Fukui Prefectural Hospital, Fukui
  - Nikko Memorial Hospital, Hokkaido
  - Dokkyo Medical University Saitama Medical Center, Saitama
- Uniwersytecki Szpital Dzieciec, Lublin, Poland
- Portugal (5):
  - CHUC - Hospital Pediatrico, Coimbra
  - Centro Hospitalar Universitaria de Lisboa Central, EPE, Lisbon
  - Centro Hospitalar Universitario Lisboa Norte, EPE, Lisbon
  - Centro Hospitalar Universitario de Porto, EPE, Porto
  - Centro Hospitalar Universitario de Sao Joao, EPE, Porto
- Romania (2):
  - Centrul de Recuperare pentru Copii dr. Nicolae Robanescu, Bucharest
  - Spitalul Clinic de Psihiatrie, Bucharest
- Almazov National Medical Research Centre, Saint Petersburg, Russia
- South Korea (7):
  - Kyungpook National University Hospital, Daegu
  - Seoul National University Bundang Hospital, Seongnam-si
  - Seoul National University Children's Hospital, Seoul
  - Severance Hospital, Seoul
  - Samsung Medical Centre, Seoul
  - Pusan National University Yangsan Hospital, Yangsan
  - Yongin Severance Hospital, Yongin-si
- Taiwan (5):
  - Kaohsiung Medical University Chung-Ho Memorial Hospital, Kaohsiung City
  - China Medical University Hospital, Taichung
  - National Taiwan University Hospital, Taipei
  - Taipei Veterans General Hospital, Taipei
  - Chang Gung Memorial Hospital Linkou Branch, Taoyuan District

IPD SHARING:
Plan to Share IPD: Undecided
Authorship of planned manuscripts for submission to medical journals shall be determined in accordance with the International Committee of Medical Journal Editors (ICMJE) Uniform Requirements for Manuscripts Submitted to Biomedical Journals (www.icmje.org).
  The physician agrees that if the physician is part of a multi-center registry, the physician shall coordinate in advance any intended disclosure of the results of the registry with Novartis Gene Therapies to ensure that the results of individual physicians are not published or presented before those of the multi-center registry, unless otherwise agreed to in writing by Novartis Gene Therapies.

REFERENCES:
- [Background] Sugarman EA, Nagan N, Zhu H, Akmaev VR, Zhou Z, Rohlfs EM, Flynn K, Hendrickson BC, Scholl T, Sirko-Osadsa DA, Allitto BA. Pan-ethnic carrier screening and prenatal diagnosis for spinal muscular atrophy: clinical laboratory analysis of >72,400 specimens. Eur J Hum Genet. 2012 Jan;20(1):27-32. doi: 10.1038/ejhg.2011.134. Epub 2011 Aug 3. PMID 21811307
- [Derived] Erbas Y, Servais L, Shieh PB, Goedeker NL, Waldrop MA, Bo R, Raju D, Benguerba K, Reyna SP, Wolff D, Finkel RS. Trach and treat: Safety and motor outcomes following onasemnogene abeparvovec in patients with spinal muscular atrophy and tracheostomies in the RESTORE registry. J Neuromuscul Dis. 2025 Nov 11:22143602251395173. doi: 10.1177/22143602251395173. Online ahead of print. PMID 41217888